CLINICAL TRIAL: NCT01700374
Title: Prepubertal Adversity Effect on Maternal Arousal, Preterm Birth and Infant Stress Response
Brief Title: Happy Mommy! Happy Baby! Study
Acronym: FAP
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 812880; P50MH099910 (NIH)
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Pregnancy; Stress, Psychological; Stress, Physiological; Maternal-fetal Relations
Keywords: pregnancy; stress, psychological; stress, physiological; maternal-fetal relations
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Salivary cortisol;
  * Blood plasma Corticotropin-releasing Hormone (CRH).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women without Prepubertal Adversity: At 8-17 weeks gestational age, 1,500 pregnant women will complete:
  * Adverse Childhood Events (ACE) Questionnaire;
  * Perceived Stress Scale (PSS);
  * A general health and demographic questionnaire.
  All women who are screened will be asked if they would be willing to allow the study team to access their delivery report.
  Women who report 0 or 1 adverse childhood experiences will be invited to continue in the study as part of the Women without Prepubertal Adversity cohort. We aim to have 125 women in this cohort.
- Women with Prepubertal Adversity: At 8-17 weeks gestational age, 1,500 pregnant women will complete:
  * Adverse Childhood Events (ACE) Questionnaire;
  * Perceived Stress Scale (PSS);
  * A general health and demographic questionnaire.
  All women who are screened will be asked if they would be willing to allow the study team to access their delivery report.
  Women who report 2 or more adverse childhood experiences will be invited to continue in the study as part of the Women without Prepubertal Adversity cohort. We aim to have 125 women in this cohort.

SUMMARY:
The purpose of this study is to determine how difficult life-events that women experienced during their childhood might affect their babies.

Women who are asked to participate in this study will fill out forms about their physical and mental health, have 3D ultrasounds of their baby's adrenal gland, have their stress responses measured and have their baby's development and stress responses assessed.

DETAILED DESCRIPTION:
The objectives of this study are to further our understanding of maternal prepubertal adversity on fetal and infant neuroendocrine development. This study utilizes 3-D ultrasound to measure fetal adrenal gland volume, a battery of psychosocial/behavioral assessments to determine the degree of maternal stress and prepubertal adversity, and an acoustic startle paradigm and Trier Social Stress Test (TSST) to assess maternal arousal. This study also utilizes an infant stress test to assess infant arousal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years;
* Able to give written informed consent;
* Between 8 to 17 weeks at time of recruitment;
* Attendance at 20 week ultrasound at a UPHS site;
* Healthy full term (35 6/7 weeks) infants;
* Fluency in written and spoken English.

Exclusion Criteria:

* Presence of a known abnormality in the present fetus, twin pregnancy or a multiple pregnancy;
* Presence of a serious medical or neurological illness, requiring treatment during pregnancy;
* Use of an antipsychotic or antidepressant medication anytime within 2 months prior to the last menstrual period;
* Drug or alcohol abuse history within previous 2 years;
* Life-time history of psychotic disorder including, schizophrenia, schizoaffective disorder; major depression with psychotic features and bipolar disorder
* Active psychiatric illness requiring treatment based upon the clinical judgement of the study psychiatrist;
* Hamilton Depression Rating Scale Score > 14;
* Suicidal ideation within the previous 6 months;
* Use of steroids drugs of antihypertensives during pregnancy as they could alter physiologic arousal;
* A history of preterm birth or history of preterm labor in the active pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women from the greater Philadelphia and surrounding areas who are ages 18 - 45 and between 8 and 17 weeks pregnant will be considered for enrollment into this study. All subjects must be physically healthy without a serious major medical illness, as well as be carrying a healthy fetus. Subjects will be recruited through fliers, advertising, and social media and may be directly approached at a University of Pennsylvania Health System (UPHS) or UPHS affiliated obstetrics and gynecology clinic. We anticipate the composition of the proposed study population to reflect the greater Philadelphia referral base. The projected composition from Philadelphia is African American 42.58%, Hispanic 8.5%, Asian 4.42%, Other 2.04% and White, not of Hispanic Origin, 42.46%.
  Additionally, we plan to include father's of the babies that are willing and able to complete the ACE questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Fetal Adrenal Size | 20 to 22 weeks gestational age
  The primary outcome variable is fetal adrenal size as measured by volume (ml) between 20 weeks and 22 weeks gestational age.

SECONDARY OUTCOMES:
Physiologic Arousal | 15 to 21 weeks gestational age and 6 to 8 weeks postpartum
  The secondary outcomes are physiologic arousal based on the maternal response to the acoustic startle paradigm or TSST plus salivary cortisol at 15-17 weeks gestational age and 6-8 weeks postpartum.
Physiologic Arousal | 6 months postpartum
  The secondary outcomes are physiologic arousal based on infant stress responses as measured by the infant behavioral assessment and salivary cortisol at 6 months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, M.D., Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - 3701 Market Street, Philadelphia, Pennsylvania
  - Helen O. Dickens Center for Women's Health, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania
  - Penn Medicine Washington Square (PMWS), Philadelphia, Pennsylvania

REFERENCES:
- [Result] Morrison KE, Epperson CN, Sammel MD, Ewing G, Podcasy JS, Hantsoo L, Kim DR, Bale TL. Preadolescent Adversity Programs a Disrupted Maternal Stress Reactivity in Humans and Mice. Biol Psychiatry. 2017 Apr 15;81(8):693-701. doi: 10.1016/j.biopsych.2016.08.027. Epub 2016 Aug 26. PMID 27776734
- See also: Program Website — http://www.med.upenn.edu/womenswellness/